CLINICAL TRIAL: NCT01374204
Title: EPILEPSY-ASSOCIATED STIGMA AND ILLNESS EXPERIENCE IN PEOPLE WITH EPILEPSY
Brief Title: Epilepsy-Associated Stigma
Acronym: EPISTIGMA
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I09004
Record Dates: First submitted 2011-06-14; First posted 2011-06-15 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Epilepsy
Keywords: Epilepsy; Stigma
MeSH Terms: conditions — Epilepsy; Social Stigma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Few data about epilepsy-associated stigma in France are available. The only study we have found showed that in France 66% of people with epilepsy felt stigmatized by their condition and are often single, compared with the other European patients interviewed (Baker et al., 2000). The purpose of this study is to assess the association between type of epilepsy (drug resistant-epilepsy and stabilized epilepsy) and perceived stigma (using the Stigma Scale) in patients recruited in the Limousin region .

DETAILED DESCRIPTION:
Epilepsy-associated stigma leads important problems in terms of public health because it can provoke significant cognitive repercussions, impairment of quality of life and it causes physical injuries and serious disabilities. These social consequences often cause more suffering for patients than seizures themselves.

This heavy medical and social burden is associated with significant economic cost in terms of care and disability. It is also noted that mortality rate is 2 to 10 times higher than the general population.

It is therefore urgent to consider both medical and social dimension of consequences of epilepsy especially in patients with uncontrolled seizures.

It is also essential to detect a potential psychiatric disorder associated with epilepsy, especially depression and anxiety which are the most prevalent psychiatric comorbidities. These disorders are often under-diagnosed that can frequently leads to an inappropriate care.

The purpose of this study is to assess the association between type of epilepsy (drug resistant-epilepsy and stabilized epilepsy) and perceived stigma (using the Stigma Scale) in patients recruited in the Limousin region .

The primary outcome will be the score of perceived stigma obtained from the Stigma Scale.

This scale estimates a score of perceived stigma for each individual and allows classifying individuals in 3 categories.

Thus, individuals who obtain a total score of 0 will be those who do not feel stigmatized. Those whose scores will be over or equal to 1will be those who feel stigmatized. Finally, respondents whose the score is equal to 3 will be considered as having a strong perception of stigma.

A positive response is characterized by threshold ≥ 1.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* diagnosed by a neurologist as suffering from drug-resistant epilepsy (all types of seizures) outpatient in Neurology service of the investigation centres
* inhabitant in the Limousin region
* having signed the informed consent
* affiliated or profiting of a social security system

Exclusion Criteria:

* patients that are deprived of their freedom
* patients with disabilities
* patients suffering from a chronic or an acute delusional disorder
* patients suffering from others handicaps

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a, descriptive and analytical study, based on a semi-directive interview among people suffering from epilepsy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-07; Primary Completion 2018-12 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
score of perceived stigma | Day one
  This scale estimates a score of perceived stigma for each individual and allows classifying individuals in 3 categories.
  Thus, individuals who obtain a total score of 0 will be those who do not feel stigmatized. Those whose scores will be over or equal to 1will be those who feel stigmatized. Finally, respondents whose the score is equal to 3 will be considered as having a strong perception of stigma.
  A positive response is characterized by threshold ≥ 1.

SECONDARY OUTCOMES:
Evaluation of the illness experience will be performed by the first section of the EMIC.
Evaluation of the representations of epilepsy (perceived causes) will be done by the second section of the EMIC

CONTACTS AND LOCATIONS:
Locations (1):
- Service de neurologie, Limoges, France